CLINICAL TRIAL: NCT04038840
Title: Imaging Synapses With [11C] UCB-J in the Human Brain
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Davidzon, Guido, M.D. (Other)
Collaborators: Weston Havens Foundation (Unknown)
Responsible Party: Principal Investigator, Jong Yoon, Associate Professor of Psychiatry and Behavioral Sciences, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 46106
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Healthy Control (HC) Participants (Experimental): Participants will undergo positron emission tomography-magnetic resonance (PET-MR) imaging using the [11C]UCB-J radiotracer
  Interventions: Drug: [11C]UCB-J radiotracer; Device: PET-MR
- Schizophrenia (SZ) Participants (Experimental): Participants will undergo positron emission tomography-magnetic resonance (PET-MR) imaging using the [11C]UCB-J radiotracer
  Interventions: Drug: [11C]UCB-J radiotracer; Device: PET-MR

INTERVENTIONS:
Drug: [11C]UCB-J radiotracer — I.V. bolus administration of up to 15 mCi (equivalent to 0.3 rems) in the antecubital vein
Device: PET-MR — Positron emission tomography and magnetic resonance imaging, with a scan duration of up to 120 minutes

SUMMARY:
The purpose of this study is to utilize the radioactive positron emission tomography (PET) tracer [11C]UCB-J to test the neural synaptic pruning hypothesis of schizophrenia. This imaging method allows for the quantification of synaptic density in the living human brain and has the unprecedented ability to directly examine the synaptic pathology underlying neuropsychiatric disease. The neural synaptic pruning hypothesis posits that a key pathogenic process of schizophrenia is the over-exuberant elimination of neural synapses during development. The confirmation of reduced synaptic density in schizophrenia as evidenced by [11C]UCB-J has the potential to lead to a number of ground-breaking clinical innovations, such as laboratory-based diagnostics and prognostics, and novel, disease-modifying treatments.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years in age
* For SZ participants:

  * On a stable medication regimen for at least two weeks prior to testing
  * A clinical diagnosis of schizophrenia, schizophreniform, or schizoaffective disorder
  * Able to complete a PET-MR scan without the use of sedation

Exclusion Criteria:

* Active substance use within three months of testing
* IQ < 70
* Major medical neurological illness or significant head trauma
* Pregnancy or breastfeeding
* Contraindication to MR scanning, including magnetic-resonance incompatible metal or hardware including pacemakers, cochlear implants, and bullets near a critical organ
* Weight > 350 lbs or a large body habitus that MR scanner cannot accommodate
* History of or current claustrophobia
* Inability to comply with basic study requirements such as following directions and punctuality
* For HC participants:

  * Presence of a first degree relative with a psychotic disorder
  * Lifetime diagnosis of major psychiatric illness
* For SZ participants:

  * Unstable psychiatric symptoms at the time of testing, e.g. acute suicidality, prominent psychosis, or behavioral dyscontrol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional differences in synaptic density between HC and SZ participants | 120 minutes (scan duration)
  Synaptic density will be quantified with the regional binding potential (BP_ND), a measure of [11C]UCB-J binding. BP_ND will be derived by using the simplified reference tissue model 2 (Wu & Carson, 2002) and the centrum semiovale as the reference region. This method has been recently utilized by other investigators in neuropsychiatric samples (Chen et al., 2018). Both exploratory voxel-wise BP_ND and region of interest (ROI) BP_ND will be compared across groups. ROIs include the striatum, dorsolateral prefrontal cortex, hippocampus, and superior temporal cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Jong H Yoon, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No
No current plan to share data

REFERENCES:
- [Background] Chong HY, Teoh SL, Wu DB, Kotirum S, Chiou CF, Chaiyakunapruk N. Global economic burden of schizophrenia: a systematic review. Neuropsychiatr Dis Treat. 2016 Feb 16;12:357-73. doi: 10.2147/NDT.S96649. eCollection 2016. PMID 26937191
- [Background] Finnema SJ, Nabulsi NB, Eid T, Detyniecki K, Lin SF, Chen MK, Dhaher R, Matuskey D, Baum E, Holden D, Spencer DD, Mercier J, Hannestad J, Huang Y, Carson RE. Imaging synaptic density in the living human brain. Sci Transl Med. 2016 Jul 20;8(348):348ra96. doi: 10.1126/scitranslmed.aaf6667. PMID 27440727
- [Background] Sekar A, Bialas AR, de Rivera H, Davis A, Hammond TR, Kamitaki N, Tooley K, Presumey J, Baum M, Van Doren V, Genovese G, Rose SA, Handsaker RE; Schizophrenia Working Group of the Psychiatric Genomics Consortium; Daly MJ, Carroll MC, Stevens B, McCarroll SA. Schizophrenia risk from complex variation of complement component 4. Nature. 2016 Feb 11;530(7589):177-83. doi: 10.1038/nature16549. Epub 2016 Jan 27. PMID 26814963
- [Background] Nabulsi NB, Mercier J, Holden D, Carre S, Najafzadeh S, Vandergeten MC, Lin SF, Deo A, Price N, Wood M, Lara-Jaime T, Montel F, Laruelle M, Carson RE, Hannestad J, Huang Y. Synthesis and Preclinical Evaluation of 11C-UCB-J as a PET Tracer for Imaging the Synaptic Vesicle Glycoprotein 2A in the Brain. J Nucl Med. 2016 May;57(5):777-84. doi: 10.2967/jnumed.115.168179. Epub 2016 Feb 4. PMID 26848175
- [Background] Feinberg I. Schizophrenia: caused by a fault in programmed synaptic elimination during adolescence? J Psychiatr Res. 1982-1983;17(4):319-34. doi: 10.1016/0022-3956(82)90038-3. PMID 7187776
- [Background] Finnema SJ, Nabulsi NB, Mercier J, Lin SF, Chen MK, Matuskey D, Gallezot JD, Henry S, Hannestad J, Huang Y, Carson RE. Kinetic evaluation and test-retest reproducibility of [11C]UCB-J, a novel radioligand for positron emission tomography imaging of synaptic vesicle glycoprotein 2A in humans. J Cereb Blood Flow Metab. 2018 Nov;38(11):2041-2052. doi: 10.1177/0271678X17724947. Epub 2017 Aug 9. PMID 28792356
- [Background] Chen MK, Mecca AP, Naganawa M, Finnema SJ, Toyonaga T, Lin SF, Najafzadeh S, Ropchan J, Lu Y, McDonald JW, Michalak HR, Nabulsi NB, Arnsten AFT, Huang Y, Carson RE, van Dyck CH. Assessing Synaptic Density in Alzheimer Disease With Synaptic Vesicle Glycoprotein 2A Positron Emission Tomographic Imaging. JAMA Neurol. 2018 Oct 1;75(10):1215-1224. doi: 10.1001/jamaneurol.2018.1836. PMID 30014145
- [Background] Wu Y, Carson RE. Noise reduction in the simplified reference tissue model for neuroreceptor functional imaging. J Cereb Blood Flow Metab. 2002 Dec;22(12):1440-52. doi: 10.1097/01.WCB.0000033967.83623.34. PMID 12468889